CLINICAL TRIAL: NCT04266652
Title: The Effect of Autogenous Tooth Roots for Lateral Alveolar Ridge Augmentation and Staged Implant Placement (A Controlled Clinical Study With Histological Assessment)
Brief Title: Using the Roots of a Non Restorable Wisdom Tooth as a Block for Augmentation of Localized Defects
Acronym: Clinical
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Lecturer Periodontology, Faculty of Dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121734
Record Dates: First submitted 2020-01-29; First posted 2020-02-12 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Augmentation
Keywords: tooth block; Dental implants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous bone block (Experimental): the monocortical block grafts were harvested from the retromolar region (i.e. linea oblique) by using of rotating (i.e. carbide burs)
  Interventions: Procedure: autogenous bone block
- Tooth block (Experimental): In the first group, a second mucoperiosteal flap was elevated to surgically remove the respective wisdom tooth. After its removal and during the same surgery, the crown was decapitated at the cemento -enamel junction using a rotating carbide bur under gentle sterile saline cooling and the exposed pulp was preserved. The separated tooth root was adapted to match the size and shape of the defect area. To improve ankylosis between the graft and the defect site, the layer of cementum at the respective downward aspects of the root was carefully removed using a diamond bur until the underlying dentin was entirely exposed
  Interventions: Procedure: tooth block

INTERVENTIONS:
Procedure: tooth block — tooth root blocks were used to increase the bone width
  Arms: Tooth block
Procedure: autogenous bone block — autogenous bone block were used to increase the bone width
  Arms: Autogenous bone block

SUMMARY:
assess and compare the efficacy and safety of autogenous tooth roots for lateral alveolar ridge augmentation with staged implant placement in comparison to autogenous bone block.

DETAILED DESCRIPTION:
A total of 14 patients in need of implant therapy and lateral ridge augmentation were allocated to parallel groups receiving either 1) healthy autogenous tooth roots (e.g. retained wisdom or impacted teeth or 2) cortical autogenous bone blocks harvested from the retromolar area. After 26 weeks of submerged healing the horizontal bone gain were assessed both clinically and radiographically. A core biopsy was taken during the implant placement to assess the histology of the newly formed bone.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for lateral ridge augmentation
2. Insufficient bone ridge width at the recipient site for implant placement
3. Sufficient bone height at the recipient site for implant placement
4. Healthy oral mucosa, at least 3 mm keratinized tissue.
5. Presence of wisdom teeth free from periapical infection.
6. Missing maxillary or mandibular tooth with moderate horizontal defect (4-8) according to cologne classification

Exclusion Criteria:

* 1) Patients are systemically free according to Modified Cornell Medical Index 2) smokers patients. 3) Pregnant or lactating women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-01-06 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic assessment of alveolar bone width following autogenous tooth roots augmentation. | 6 months postoperatively

SECONDARY OUTCOMES:
Histological analysis of remodeled autogenous bone roots 4 months following horizontal ridge augmentation. Histological analysis of remodeled autogenous bone roots 4 months following horizontal ridge augmentation. | 6 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt